CLINICAL TRIAL: NCT07169279
Title: Phase 2b, Randomized, Double-Blind, Placebo-Controlled Clinical Trial, Preceded by a Single Ascending Dose Portion and a Phase 2 Open-Label Portion, to Evaluate the Safety and Efficacy of Oral Infigratinib in Infants and Young Children With Achondroplasia
Brief Title: Interventional Study of Infigratinib in Children < 3 Years Old With Achondroplasia (ACH)
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: QED Therapeutics, a BridgeBio company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: QBGJ398-204
Record Dates: First submitted 2025-06-23; First posted 2025-09-11 (Actual); Last update posted 2025-12-15 (Actual); Status verified 2025-12

CONDITIONS: Achondroplasia
Keywords: skeletal dysplasia; endochondral ossification; achondroplasia; ACH; Shortened proximal limbs; fibroblast growth factor receptor 3; FGFR3; encodhondral bone formation; disproportionate short stature; quality of life; dwarfism; bone diseases; musculoskeletal diseases; osteochondrodysplasia; functional abilities; annualized growth velocity; annualized height velocity; growth; growth disorder; congenital; AHV; AGV; infant and toddler
MeSH Terms: conditions — Achondroplasia; Mucopolysaccharidosis IV; Dwarfism; Bone Diseases; Musculoskeletal Diseases; Osteochondrodysplasias; Growth Disorders | interventions — Administration, Oral; infigratinib

STUDY DESIGN:
Intervention Model Description: This study comprises 4 portions: a Single Ascending Dose (SAD) portion and open-label Phase 2 portion to evaluate safety and PK and select a dose level for Phase 2b; a placebo-controlled Phase 2b portion, to assess safety and efficacy at the selected dose level; and an open-label extension portion to evaluate safety and efficacy in children < 3 years old who have completed the Phase 2 or Phase 2b portion of the study.
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (15):
- SAD Cohort 1 infigratinib (2 to less than 3 years old) (Experimental): Single Ascending Dose Escalation and PK Portion
  Interventions: Drug: Infigratinib is provided as a single dose of minitablets for oral administration
- SAD Cohort 2 infigratinib (1 to less than 2 years old) (Experimental): Single Ascending Dose Escalation and PK Portion
  Interventions: Drug: Infigratinib is provided as a single dose of minitablets for oral administration
- SAD Cohort 3 infigratinib (6 months to less than 1 year old) (Experimental): Single Ascending Dose Escalation and PK Portion
  Interventions: Drug: Infigratinib is provided as a single dose of minitablets for oral administration
- SAD Cohort 4 infigratinib (0 to less than 6 months old) (Experimental): Single Ascending Dose Escalation and PK Portion
  Interventions: Drug: Infigratinib is provided as a single dose of minitablets for oral administration
- Phase 2 Cohort 1 infigratinib (2 to less than 3 years old) (Experimental): Open-label Safety and PK Portion
  Interventions: Drug: Infigratinib is provided as sprinkle capsules for daily oral administration
- Phase 2 Cohort 2 infigratinib (1 to less than 2 years old) (Experimental): Open-label Safety and PK Portion
  Interventions: Drug: Infigratinib is provided as sprinkle capsules for daily oral administration
- Phase 2 Cohort 3 infigratinib (6 months to less than 1 year old) (Experimental): Open-label Safety and PK Portion
  Interventions: Drug: Infigratinib is provided as sprinkle capsules for daily oral administration
- Phase 2 Cohort 4 infigratinib (0 to less than 6 months) (Experimental): Open-label Safety and PK Portion
  Interventions: Drug: Infigratinib is provided as sprinkle capsules for daily oral administration
- Phase 2B Cohort 1 infigratinib (2 to less than 3 years old) (Experimental): Randomized Safety and Efficacy Portion
  Interventions: Drug: Infigratinib or placebo comparator is provided as sprinkle capsules for daily oral administration
- Phase 2B Cohort 2 infigratinib (6 months to less than 2 years old) (Experimental): Randomized Safety and Efficacy Portion
  Interventions: Drug: Infigratinib or placebo comparator is provided as sprinkle capsules for daily oral administration
- Phase 2B Cohort 3 infigratinib (0 to less than 6 months old) (Experimental): Randomized Safety and Efficacy Portion
  Interventions: Drug: Infigratinib or placebo comparator is provided as sprinkle capsules for daily oral administration
- Open- label Extension infigratinib (0 months to 3 years [+6 months old]) (Experimental): Open-label extension portion continuing to assess safety and efficacy in children until they reach 3 years old (+6 months)
  Interventions: Drug: Infigratinib is provided as sprinkle capsules for daily oral administration
- Phase 2B Cohort 1 Placebo (2 to less than 3 years old) (Placebo Comparator): Randomized Safety and Efficacy study
  Interventions: Drug: Infigratinib or placebo comparator is provided as sprinkle capsules for daily oral administration
- Phase 2B Cohort 2 placebo (6 months to less than 2 years old) (Placebo Comparator): Randomized Safety and Efficacy study
  Interventions: Drug: Infigratinib or placebo comparator is provided as sprinkle capsules for daily oral administration
- Phase 2B Cohort 3 Placebo (0 to less than 6 months old) (Placebo Comparator): Randomized Safety and Efficacy study
  Interventions: Drug: Infigratinib or placebo comparator is provided as sprinkle capsules for daily oral administration

INTERVENTIONS:
Drug: Infigratinib is provided as a single dose of minitablets for oral administration — * The initial cohort dose of infigratinib will begin at the protocol-specified starting dose, with subsequent cohort escalation based on protocol specific criteria.
  * The target dose is the dose that will provide similar exposure to the dose of 0.25 mg/kg/day in participants 3 years old and older.
  * The dose and number of minitablets will be calculated based on individual participant age and weight.
  Arms: SAD Cohort 1 infigratinib (2 to less than 3 years old); SAD Cohort 2 infigratinib (1 to less than 2 years old); SAD Cohort 3 infigratinib (6 months to less than 1 year old); SAD Cohort 4 infigratinib (0 to less than 6 months old)
Drug: Infigratinib is provided as sprinkle capsules for daily oral administration — * The cohort dose of infigratinib will be the dose identified in the Single Ascending Dose portion for the age group.
  * The dose and number of sprinkle capsules/day will be calculated based on individual participant age and weight. Doses will be adjusted based on age and weight changes approximately every 3 months.
  Arms: Phase 2 Cohort 1 infigratinib (2 to less than 3 years old); Phase 2 Cohort 2 infigratinib (1 to less than 2 years old); Phase 2 Cohort 3 infigratinib (6 months to less than 1 year old); Phase 2 Cohort 4 infigratinib (0 to less than 6 months)
Drug: Infigratinib or placebo comparator is provided as sprinkle capsules for daily oral administration — * The cohort dose of infigratinib or placebo will be the dose confirmed in the Phase 2 portion for the age group.
  * The dose and number of sprinkle capsules/day will be calculated based on individual participant age and weight. Doses will be adjusted based on age and weight changes approximately every 3 months.
  Arms: Phase 2B Cohort 1 Placebo (2 to less than 3 years old); Phase 2B Cohort 1 infigratinib (2 to less than 3 years old); Phase 2B Cohort 2 infigratinib (6 months to less than 2 years old); Phase 2B Cohort 2 placebo (6 months to less than 2 years old); Phase 2B Cohort 3 Placebo (0 to less than 6 months old); Phase 2B Cohort 3 infigratinib (0 to less than 6 months old)
Drug: Infigratinib is provided as sprinkle capsules for daily oral administration — * The dose of infigratinib will be the dose confirmed in the Phase 2 portion and used in the Phase 2b portion for the age group.
  * The dose and number of sprinkle capsules/day will be calculated based on individual participant age and weight. Doses will be adjusted based on age and weight changes approximately every 3 months for the first year and every 6 months thereafter.
  Arms: Open- label Extension infigratinib (0 months to 3 years [+6 months old])

SUMMARY:
This is a Phase 2, multicenter, randomized, placebo-controlled study to evaluate the safety and efficacy of infigratinib in participants < 3 years old with ACH. The purposes of the SAD and Phase 2 portions are to identify and confirm the dose of infigratinib to be used in the Phase 2b portion, based on safety and PK. The purpose of the Phase 2b, placebo-controlled portion is to evaluate the safety and efficacy of infigratinib in children < 3 years old with ACH at the selected dose.

DETAILED DESCRIPTION:
PROPEL Infant & Toddler (I&T) is a Phase 2, multicenter, randomized, placebo-controlled study that comprises 4 portions: the single ascending dose (SAD) portion (open-label), the Phase 2 portion (open-label), the Phase 2b portion (placebo-controlled), and an Extension Portion (open-label). The study will evaluate children with ACH < 3 years old being administered oral infigratinib.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of ACH confirmed by genetic testing. If prospective participants had prior genetic testing, the diagnosis must be confirmed by a report from a certified laboratory, documenting the specific mutation.
* Age 0 to 32 months (2 years and 8 months) at screening.
* Signed informed consent, which must be obtained from each participant's parent(s) or legal guardian.
* Parent(s)/Guardian(s) willing and able to attend all study visits and comply with all study requirements.
* Parent(s)/Guardian(s) willing and able to comply with the routine care of the study participants according to local guidance for the management of infants and young children with ACH.
* Able to swallow age-appropriate oral medication.
* In participants <1 year old, be compliant with recommended vitamin D supplementation of 5 10 μg/day or higher (or as recommended by country specific guidelines).

Exclusion Criteria:

* Participants who have hypochondroplasia or diagnosis of genetic condition other than ACH, or any clinical condition that can affect growth.
* Gestational age at birth <37 weeks and/or birth weight <2500 grams.
* Gastroesophageal reflux disease requiring prolonged treatment (>1 week) with prohibited medications.
* Evidence of cervicomedullary compression, as defined by an Achondroplasia Foramen Magnum Score (AFMS) 4, symptomatic or asymptomatic, diagnosed during MRI done at screening or a previous MRI done at any time if the participant had not undergone decompression surgery.
* History of fracture of a long bone or spine within 6 months prior to screening.
* Any other significant concurrent disease or condition that, in the view of the investigator and/or sponsor, would confound assessment of efficacy or safety of infigratinib and/or would require treatment with a prohibited medication (per protocol), and/or would place the participant at high risk for poor treatment compliance or for failure to complete the study.
* Having received or planning to receive treatment with any other investigational or approved product for the treatment of ACH or short stature, including (but not limited to) r-hGH, IGF-1, CNP analog, FGF ligand trap, or treatment targeting FGFR inhibition at any time.
* Regular long-term (>3 weeks; more than twice/year) treatment with supraphysiologic doses of glucocorticoid therapy (ie, >15 mg/m2/day of hydrocortisone or equivalent) or treatment with glucocorticoids at anti-inflammatory doses (for over 3 weeks within 6 months of the screening visit. NOTE: Low-dose topical, inhaled, or intranasal corticosteroids are acceptable.
* Significant abnormality in screening laboratory results,
* Allergy or hypersensitivity to any components of the study drug.

Ages: 0 Years to 32 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 77 (Estimated)
Dates: Start 2025-11-19 (Actual); Primary Completion 2032-03 (Estimated); Study Completion 2032-03 (Estimated)

PRIMARY OUTCOMES:
Single Ascending Dose Portion: Identify the dose of infigratinib to be used in each age cohort of the Phase 2 potion of the study (by assessing safety and PK of infigratinib and its active metabolites) | 2 weeks
Phase 2 Portion: Confirm the doses to be used in each age cohort in the Phase 2b portion of the study (by assessing safety and PK of infigratinib and its active metabolites). | 52 weeks
Phase 2b Portion: Evaluate the safety and efficacy of infigratinib in infants and children < 3 years old with ACH (by assessing AE's & SAE's) | 52 weeks
Extension Portion: Evaluate the safety and efficacy of infigratinib in participants who completed the Phase 2 or Phase 2b portion of the study until they have reached 3 years old (+6 months) (by assessing AE's and SAE's) | 3 years and 6 months

SECONDARY OUTCOMES:
Phase 2: Evaluate the safety of oral daily doses of infigratinib (by assessing AEs and SAEs) | 52 weeks
Phase 2: Evaluate changes in indicators of growth (by assessing change from BL in body length z-score at Week 52 in relation to ACH tables) | 52 weeks
Phase 2: Evaluate changes in indicators of body proportions (by assessing change from BL to Week 52 in upper-to-lower body segment ratio and head circumference/body length ratio) | 52 weeks
Phase 2: Change from BL in Health-related Quality of Life (HRQoL) (as assessed by Infant and Toddler Quality of Life Inventory [ITQoL] tool) | 52 weeks
Phase 2: Milestone Development of motor skills (assessed with development milestone charts) | 52 weeks
Phase 2: Milestone Development of language skills (assessed with development milestone charts) | 52 weeks
Phase 2: Milestone Development of personal-social skills (assessed with development milestone charts) | 52 weeks
Phase 2: Skull and brain morphology (as assessed using MRI) | 52 weeks
Phase 2: Age at closure of cranial structures (as assessed by physical examination) | 52 weeks
Phase 2: Age at closure of fontanelles (as assessed by physical examination) | 52 weeks
Phase 2: Incidence of surgical interventions (i.e., cervical decompression, adenotonsillectomy etc) | 52 weeks
Phase 2: Incidence and severity of sleep apnea (as assessed by polysomnography) | 52 weeks
Phase 2: Bone morphology (as assessed using x-rays) | 52 weeks
Phase 2b: Evaluate the pharmacokinetic (PK) profile of infigratinib and its metabolites (by assessing the PK of infigratinib and its active metabolites) | 52 weeks
Phase 2b: Change from BL in Health-related Quality of Life (HRQoL) (as assessed by Infant and Toddler Quality of Life Inventory [ITQoL] tool) | 52 weeks
Phase 2b: Evaluate the safety of oral daily doses of infigratinib (by assessing AEs and SAEs) | 52 weeks
Phase 2b: Evaluate changes in indicators of growth (by assessing change from BL in body length z-score at Week 52 in relation to ACH tables) | 52 weeks
Phase 2b: Evaluate changes in indicators of body proportions (by assessing change from BL to Week 52 in upper-to-lower body segment ratio and head circumference/body length ratio) | 52 weeks
Phase 2b: Milestone Development of motor skills (assessed with development milestone charts) | 52 weeks
Phase 2b: Milestone development of language skills (assessed with development milestone charts) | 52 weeks
Phase 2b: Milestone development of personal-social skills (assessed with development milestone charts) | 52 weeks
Phase 2b: Skull and brain morphology (as assessed using MRI) | 52 weeks
Phase 2b: Age at closure of cranial structures (as assessed by physical examination) | 52 weeks
Phase 2b: Age at closure of fontanelles (as assessed by physical examination) | 52 weeks
Phase 2b: Incidence of surgical interventions (i.e., cervical decompression, adenotonsillectomy etc) | 52 weeks
Phase 2b: Incidence and severity of sleep apnea (as assessed by polysomnography) | 52 weeks
Phase 2b: Bone morphology (as assessed using x-rays) | 52 weeks
Extension Phase: Evaluate the safety of oral daily doses of infigratinib (by assessing AEs and SAEs) | Until they have reached 3 years old (+6 months)
Extension Phase: Change from BL in body length Z-score | Until they have reached 3 years old (+6 months)
Extension Phase: Change from BL in upper to lower body segment ratio (cm) | Until they have reached 3 years old (+6 months)
Extension Phase: Change from BL in head circumference body length ratio | Until they have reached 3 years old (+6 months)
Extension Phase: Milestone development of social/emotional skills (assessed with development milestone charts) | Until they have reached 3 years old (+6 months)
Extension Phase: Milestone development of language communication skills (assessed with development milestone charts) | Until they have reached 3 years old (+6 months)
Extension Phase: Milestone development of cognitive skills (assessed with development milestone charts) | Until they have reached 3 years old (+6 months)
Extension Phase: Milestone development of movement/physical development skills (assessed with development milestone charts) | Until they have reached 3 years old (+6 months)
Extension Phase: Age at closure of cranial structures (as assessed by physical examination) | Until they have reached 3 years old (+6 months)
Extension Phase: Age at closure of fontanelles (as assessed by physical examination) | Until they have reached 3 years old (+6 months)
Extension Phase: Incidence of surgical interventions (i.e., cervical decompression, adenotonsillectomy etc) | Until they have reached 3 years old (+6 months)
Extension Phase: Bone morphology (as assessed using x-rays) | Until they have reached 3 years old (+6 months)

CONTACTS AND LOCATIONS:
Locations (13):
- United States (3):
  - UCSF Benioff Children's Hospital, Oakland, California
  - Johns Hopkins University, Baltimore, Maryland
  - University of Wisconsin Madison - Waisman Center Bone Dysplasia Clinic, Madison, Wisconsin
- Murdoch Children's Research Institute, Parkville, Victoria, Australia
- Canada (2):
  - Children's Hospital of Eastern Ontario Research Institute, Ottawa, Ontario
  - Université de Montréal - Centre Hospitalier Universitaire Sainte-Justine, Montreal, Quebec
- Paediatric Clinical Research Unit at Oslo University Hospital, Oslo, Norway
- KK Women's and Children's Hospital, Singapore, Singapore
- Unidad de Cirugia Artroscopica (UCA), Vitoria-Gasteiz, Spain
- United Kingdom (4):
  - NHS Greater Glasgow and Clyde, Glasgow
  - Guy's and Saint Thomas' NHS Foundation Trust, London
  - Manchester University NHS Foundation Trust, Manchester
  - Sheffield Children's NHS Foundation Trust, Sheffield

IPD SHARING:
Plan to Share IPD: No